CLINICAL TRIAL: NCT05761964
Title: Harmony & Health: Feasibility of a Movement Intervention to Improve Psychosocial Wellbeing in Black Adults in Northeast Texas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Duncan Family Institute (DFI) Seed Funding Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0793; NCI-2023-01856 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-23; First posted 2023-03-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Psychological
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health and Harmony (Experimental): Participants will take part in a program combining yoga practices and Christian spirituality.
  Interventions: Behavioral: Harmony & Health; Behavioral: Health Education
- Health Education (Control) (Other): Participants will take part in a series of health education sessions.
  Interventions: Behavioral: Harmony & Health; Behavioral: Health Education

INTERVENTIONS:
Behavioral: Harmony & Health — Participants will attend group in-person sessions 2 times each week for 8 weeks. The session will be 45 minutes long. In each session, there will be an introduction, 30 minutes of gentle yoga-based poses and breathing exercises, and then 10 minutes of guided relaxation and scripture meditation. Participants will be asked to complete at-home stretching practices 2 times each week for the 8 week intervention period. Participants will also be asked to complete weekly logs to self-monitor their physical activity.
Behavioral: Health Education — Participants will attend group in-person health education sessions 2 times each week for 8 weeks. The sessions will be 45 minutes long and will include discussions of disease prevention and other health and wellbeing topics.

SUMMARY:
To test the feasibility and acceptability of a program that combines yoga practices and Christian spirituality (called Harmony & Health) amongst insufficiently active Black adults.

DETAILED DESCRIPTION:
Objectives

Primary Objective:

The primary objective of this 2-arm randomized controlled pilot study is to test the feasibility and acceptability of HH in Black adults residing in rural areas surrounding Tyler in Northeast Texas. Black adults who are insufficiently active will be randomized to the HH intervention or an attention control group. We hypothesize that we will meet our recruitment goal of 50 participants over 5 months, ≥80% of participants will be retained at post-intervention and follow up, and ≥80% will adhere to sessions.

Secondary Objectives:

The secondary objectives of this study are:

2.a. To explore the effects of HH on sitting time and LPA in Black adults who are insufficiently active. Participants will complete assessments at baseline (week 0), post-intervention (week 9), and follow-up (week 24), and changes in measured sitting time and LPA from week 0 to 9 will be assessed.

2.b. To evaluate acceptability of the intervention and assessment protocols via in-depth interviews. After follow-up, we will conduct interviews with community partners (n=2), delivery agents (n=2), and participants (n=16) to assess acceptance and refine training and implementation protocols in preparation for a future large-scale randomized controlled efficacy trial.

ELIGIBILITY:
Inclusion criteria:

1. Men and women ≥18 years of age
2. Self-identify as Black or African American
3. Able to read, speak, and write in English
4. Primary residence in the Northeast Texas area (Public Health Region 4/5N)
5. Insufficiently active (self-report <75 minutes/week of physical activity)
6. Sedentary (self-report ≥6 hours/day of sitting time)
7. Body mass index [BMI] ≥25 kg/m2
8. Able to pass the Physical Activity Readiness Questionnaire (PARQ) or provide physician's clearance to participate
9. Able to provide written informed consent without assistance

Exclusion criteria:

1. <18 years of age
2. Do not self-identify as Black or African American
3. Unable to read, speak, and write in English
4. Primary residence falls outside of the Northeast Texas area or Public Health Region 4/5N
5. Physically active or self-report doing ≥75 minutes/week of physical activity
6. Not sedentary or self-report <6 hours/day of sitting time
7. BMI <25.0 kg/m2
8. Absolute contraindications to unassisted physical activity based on the PARQ (e.g., acute MI, orthopedic and musculoskeletal limitations)
9. Planning to move from the Northeast Texas during the 6 month study period
10. Pregnant or planning to become pregnant during the 6 month study period
11. Currently participating in another program to increase physical activity, reduce sedentary behavior, or manage weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the intervention: Recruitment and retention | through study completion; an average of 1 year.
  Rates of study eligibility, recruitment, and retention will be assessed. We will maintain detailed information during the recruitment process regarding the number of church members interested, eligible, ineligible and reasons for ineligibility, and enrolled. To assess feasibility, we will calculate the rates of study eligibility, recruitment, and retention, along with their 90% confidence intervals (CIs). Participant feedback will be summarized using means and standard deviations along with graphical display (e.g., box plots). Recruitment success, i.e., feasibility will be achieved if ≥50% of eligible participants enrolls in the study. Retention success will be achieved if ≥80% participants complete the post-intervention and follow-up assessments.
Feasibility and acceptability of the intervention: Program satisfaction | through study completion; an average of 1 year.
  Following the follow-up data collection time point, we will conduct individual interviews with a subsample of participants (~16 participants). Interview questions will address participants' overall reactions to and satisfaction with the mind-body intervention, perceived impact on social support, motivation, and self-efficacy for increase physical activity and well-being. Positive satisfaction, i.e., successful feasibility, will be achieved when participants consistently and repeatedly, through subsequent interviews, endorse satisfaction with the program through use of positive language when describing their feelings toward the program. Interviews will be conducted by the PI or trained member of the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Scherezade Mama, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://mdanderson.org